CLINICAL TRIAL: NCT04448353
Title: Carotid Risk Prediction (CRISP) Consortium
Acronym: CRISP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Elucid Bioimaging Inc. (Industry)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Other Study IDs: CRISP
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-06

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Development / training: Selected by stratified partitioning
  Interventions: Diagnostic Test: vascuCAP
- Sequestered / test: Selected by stratified partitioning
  Interventions: Diagnostic Test: vascuCAP

INTERVENTIONS:
Diagnostic Test: vascuCAP — adverse event and phenotype classification model

SUMMARY:
Develop adverse event prediction and plaque phenotype classification models for patients with known or suspected carotid artery disease.

DETAILED DESCRIPTION:
Develop adverse event prediction and plaque phenotype classification models using plaque morphology and composition assessment of CTA which has been validated by histology, applied to representative cohort of patients. Generalizability of models is enhanced by using validated rather than only raw image inputs. Demographic, clinical, and outcome data is collected for enrolled patients as well as information on events and interventions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have two (or more) neck CTAs at least 6 months apart of sufficient quality as documented in the vascuCAP Reading Manual.
* Atherosclerotic plaque must be visualized within the carotid artery.

Exclusion Criteria:

* Subjects without visible plaque within the carotid artery
* Subject with insufficient CTA image quality (defined strictly as documented in the vascuCAP Reading Manual)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All-comers, design, adjusted for demographic factors
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse outcome model performance | 2 years
  Develop adverse event model for major adverse neurological events (MANE) prediction on large retrospective cohort (and enable a prospective collection subsequent to this study). Consistent with this primary endpoint is the evaluation of all imaging-derived data that has a bearing on the diagnosis and prognosis of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Brajesh K. Lal, MD, Principal Investigator — University of Maryland, College Park
Locations (5):
- United States (5):
  - Baltimore VA Medical Center, Baltimore, Maryland
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Weill Cornell Medicine (Affiliated with New York Presbyterian Hospital), New York, New York
  - University Hospital Harrington (Affiliated with Case Western Reserve University), Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lal BK, Khan AA, Kashyap VS, Chrencik MT, Gupta A, King AH, Patel JB, Martinez-Delcid J, Uceda D, Desikan S, Sikdar S, Sorkin JD, Buckler A. Computed tomography angiographic biomarkers help identify vulnerable carotid artery plaque. J Vasc Surg. 2022 Apr;75(4):1311-1322.e3. doi: 10.1016/j.jvs.2021.10.056. Epub 2021 Nov 15. PMID 34793923